CLINICAL TRIAL: NCT04033328
Title: An Open-Label Phase 1b Study of ORIC-101 in Combination With Enzalutamide in Patients With Metastatic Prostate Cancer Progressing on Enzalutamide
Brief Title: Study of ORIC-101 in Combination With Enzalutamide
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IND Withdrawn
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORIC-101-02
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: Modified interval 3+3 dose escalation design, followed by dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): ORIC-101 dosed orally, once per day in combination with enzalutamide (160 mg) of each 28-day cycle.
  Interventions: Drug: ORIC-101; Drug: enzalutamide 40 MG oral capsule [Xtandi]
- Dose Expansion (Experimental): RP2D dose
  Interventions: Drug: ORIC-101; Drug: enzalutamide 40 MG oral capsule [Xtandi]

INTERVENTIONS:
Drug: ORIC-101 — ORIC-101 once daily in each 28-day cycle
Drug: enzalutamide 40 MG oral capsule [Xtandi] — 160 mg once daily in each 28-day cycle

SUMMARY:
The purpose of this study is to establish the recommended phase 2 dose (RP2D), safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of ORIC-101 in combination with enzalutamide (Xtandi®) when administered to patients with metastatic prostate cancer progressing on enzalutamide.

DETAILED DESCRIPTION:
ORIC-101 is a small molecule GR antagonist being developed for the treatment of patients with solid tumor malignancies. Mechanistically, ORIC-101 inhibits GR transcriptional activity and blocks the pro-survival signals mediated by the activated nuclear receptor.

This is an open-label, single arm, multicenter, dose escalation followed by dose expansion study to assess the safety and preliminary antitumor activity of ORIC-101 in combination with enzalutamide in patients progressing on enzalutamide. Patients deemed eligible will receive treatment with ORIC-101 in addition to continuing their current enzalutamide therapy.

Escalating dose levels of ORIC-101 will be administered orally, once daily in combination with enzalutamide 160 mg. Parallel enrollment for assessment of PK/PD modulation in up to 3 additional patients presenting with tumors expressing high levels of GR (GR-high) may be performed at each dose level after the dose level has cleared the initial dose-limiting toxicity evaluation period; these additional patients may serve as supplemental patients for selection of the maximum tolerated dose and/or RP2D.

Dose expansion will further evaluate the safety and preliminary antitumor activity of ORIC-101 in patients presenting with different levels of GR expressing-tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Metastatic prostate cancer currently being treated with enzalutamide (Xtandi®) 160 mg once daily plus surgical or ongoing chemical castration, with baseline testosterone level <50 ng/dL
* Must have been on treatment with enzalutamide for at least 3 months prior to documented evidence of PSA progression defined as per PCWG3: minimum of 2 rising values (3 measurements) obtained a minimum of one week apart with the latest result being at least 2.0 ng/mL (or 1.0 ng/mL if PSA rise is the only indication of progression)
* Agreement and ability to undergo on-study core biopsies, as follows, through a procedure that is deemed to be clinically feasible and not carry significant risk:

  * one pre-treatment tumor biopsy obtained while on treatment with enzalutamide prior to enrollment on this study; and
  * one post-treatment tumor biopsy during Cycle 2
  * one end of treatment tumor biopsy (optional)
* ECOG performance status 0 or 1
* Life expectancy of at least 3 months
* Adequate organ function as defined by the following criteria:

  * ANC ≥1500 cells/mm3 (1.5 × 103 cells/mm3)
  * Platelets ≥100,000 /µL (100 × 109 /L)
  * Hemoglobin ≥9.0 g/dL (90 g/L)
  * AST (SGOT) or ALT (SGPT) ≤2.5 × ULN, ≤5.0 × ULN for patients with liver metastases
  * Bilirubin ≤1.5 × ULN; patients with a known history of Gilbert's syndrome and/or isolated elevations of indirect bilirubin are eligible
  * QTcF ≤480 msec
* Capable of giving signed informed consent

Exclusion Criteria:

* No intervening therapy between enzalutamide treatment and enrollment on this study
* Any other active malignancy, with the exception of adequately treated non-melanoma skin cancer, adequately treated superficial bladder cancer, stage 1 or 2 solid tumor malignancies without evidence of disease, or other solid tumors curatively treated with no evidence of disease for ≥5 years from enrollment
* Current treatment on another therapeutic clinical trial
* Prior or current treatment with ORIC-101 or any other GR antagonist (eg, CORT-125281, mifepristone, relacorilant)
* Prior chemotherapy in the metastatic castration-resistant prostate cancer setting
* Prior treatment with a second-generation AR modulator (eg, apalutamide, abiraterone, darolutamide)
* History of Cushing's syndrome or adrenal insufficiency
* History or presence of CNS metastases
* History of seizures or condition that may predispose to seizures
* Current (at C1D1) or requirement for chronic use of systemic corticosteroids with the exception of inhaled, topical, intraocular, intranasal, or intraarticular corticosteroids
* Current (within 10 days prior to first dose of ORIC-101) or expected on-study treatment with specified strong CYP3A4 inhibitors or inducers
* Receiving any other anticancer therapy, including radiotherapy within 21 days prior to C1D1. Patients must have recovered from all toxicities from prior anticancer therapies and/or radiotherapy
* Major surgery within 21 days prior to C1D1 or incomplete recovery from adverse effects resulting from such procedure
* Known human immunodeficiency virus (HIV) infection, unless patient is healthy and has a low risk of AIDS-related outcomes
* Active Hepatitis B or C infection
* Any other condition or circumstance (eg, clinical, psychological, familial, sociological, inability to swallow oral study drug) that, in the opinion of the investigator, may interfere with protocol compliance or contraindicates participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 12 months
  RP2D as determined by 3+3 dose escalation design
PSA Response Rate | 36 months
  ≥50% decline from baseline at 8 weeks per Prostate Cancer Working Group 3 (PCWG3) criteria
PSA Progression | 36 months
  From study start until PCWG3 criteria is met
Number of Participants with Adverse Events | 36 months
  Safety and tolerability of ORIC-101 in combination with enzalutamide
Number of Participants with Abnormal Laboratory Values | 36 months
  Safety and tolerability of ORIC-101 in combination with enzalutamide
Number of Participants with Abnormal 12-lead ECG | 36 months
  Safety and tolerability of ORIC-101 in combination with enzalutamide
Number of Participants with Abnormal Vital Signs | 36 months
  Safety and tolerability of ORIC-101 in combination with enzalutamide

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 Days
  PK of ORIC-101 in combination with enzalutamide
Minimum plasma concentration (Cmin) | 36 months
  PK of ORIC-101 in combination with enzalutamide
Time of maximum observed concentration (Tmax) | 28 Days
  PK of ORIC-101 in combination with enzalutamide
Area under the curve (AUC(0-24)) | 28 Days
  PK of ORIC-101 in combination with enzalutamide
Elimination half-life (T1/2) | 28 Days
  PK of ORIC-101 in combination with enzalutamide
Circulating tumor cells (CTCs) conversion | 36 months
  ≥5 cells/7.5 mL of blood to 0 (zero) (CTC0), as well as from unfavorable (≥5 cells/7.5 mL of blood) to favorable (<5 cells/7.5 mL of blood)
Objective response rate (ORR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and PCWG3 criteria
Duration of response (DOR) | 36 months
  Radiographic progression using RECIST v1.1
Progression-free survival (PFS) | 36 months
  Time from first dose to first documentation of radiographic progression or death
Overall survival (OS) | 36 months
  Time from first dose to death
Number of Participants with GR Expression by IHC | 36 months
  Level of GR expression by IHC in tumor tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S. Multani, MD, Study Director — ORIC Pharmaceuticals
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Abida W, Hahn AW, Shore N, Agarwal N, Sieber P, Smith MR, Dorff T, Monk P, Rettig M, Patel R, Page A, Duff M, Xu R, Wang J, Barkund S, Pankov A, Wang A, Junttila MR, Multani PS, Daemen A, Chow Maneval E, Logothetis CJ, Morris MJ. Phase I Study of ORIC-101, a Glucocorticoid Receptor Antagonist, in Combination with Enzalutamide in Patients with Metastatic Castration-resistant Prostate Cancer Progressing on Enzalutamide. Clin Cancer Res. 2024 Mar 15;30(6):1111-1120. doi: 10.1158/1078-0432.CCR-23-3508. PMID 38226958